CLINICAL TRIAL: NCT05296135
Title: Predicting Immunotherapy Efficacy from Analysis of Pre-treatment Tumor Biopsies, Head and Neck Squamous Cell Cancer, Study 2
Brief Title: Predicting Immunotherapy Efficacy in Head and Neck Squamous Cell Cancer
Acronym: PREDAPT-HNSCC2
Status: Withdrawn | Type: Observational
Why Stopped: No patients were recruited or enrolled in this study.
Sponsor: Cofactor Genomics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PREDAPT-HNSCC-2
Record Dates: First submitted 2022-03-07; First posted 2022-03-25 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Main Cohort
  Interventions: Diagnostic Test: OncoPrism-HNSCC™

INTERVENTIONS:
Diagnostic Test: OncoPrism-HNSCC™ — OncoPrism-HNSCC™ is a new approach to characterizing the immune component of pre-treatment tumor tissue.

SUMMARY:
This study will investigate the clinical validity and clinical utility of the OncoPrism-HNSCC (Head and Neck Squamous Cell Carcinoma) test.

DETAILED DESCRIPTION:
Patient outcomes would be improved if the available molecular diagnostics for predicting response to immunotherapy, namely PD-L1 immunohistochemistry (IHC) scoring, had greater accuracy in predicting tumor response. While PD-L1 expression in tumor specimens roughly correlates with benefit from immunotherapy, the predictive value of PD-L1 expression is low.

To address these weaknesses, new diagnostic methods are needed to accurately predict patient benefit from immunotherapy. As part of this effort, the investigators propose to evaluate the Cofactor OncoPrism-HNSCC™ assay.

The OncoPrism-HNSCC test is a qualitative Next Generation Sequencing (NGS)-based messenger ribonucleic acid (mRNA) gene expression profiling test system intended for use with FFPE tumor tissue to identify and analyze onco-immune phenotype molecular signatures and generate a prognostic score and classifier for previously diagnosed patients considered for treatment with immunotherapy.

Given a pre-treatment FFPE tumor specimen, OncoPrism-HNSCC™ (OP) Laboratory Derived Test (LDT) reports on a OncoPrism Score (OPS) for each patient. The test results assign patients to 1 of 4 intervals depending on the patient's OPS, with higher scores, and higher intervals correlating to higher immunotherapy efficacy. This study will measure the clinical outcomes of patients according to each interval.

The investigators hypothesize that the results from this study will show that the OncoPrism-HNSCC test is prognostic of the efficacy of immunotherapy. Specifically, the investigators hypothesize that clinical outcomes will be better for those patients who are assigned to higher intervals, according to the test.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have been diagnosed with recurrent or metastatic HNSCC.
2. Subject must have received, or be scheduled to receive, at least one dose of FDA approved anti-PD-1/PD-L1 immunotherapy for treatment of their cancer.
3. Subject must have had, or will have, a tumor biopsy prior to treatment with anti-PD-1/PD-L1 immunotherapy.
4. Subject must have a RECIST determination of PD-L1/PD-1 inhibitor-treatment by imaging or clinical assessment.
5. Willing to provide electronic informed consent per IRB-approved protocol.
6. Able to speak, read, and comprehend English or Spanish fluently.
7. Subject is 18 years of age or older.
8. Subjects must have sufficient tissue available to fulfill the specimen requirements of the study, as defined in the Specimens to be Collected section of protocol.

Exclusion Criteria:

1. Subject shall not have received immunotherapy in combination with other therapy modality such as radiation therapy, platinum-based chemotherapy, or a taxane.
2. Subject shall not have received immunotherapy outside of FDA approved use as of the date of this protocol.
3. Subject shall not have inability or unwillingness to provide informed consent.
4. Subject shall not have other cancers than listed above (other histologies).
5. Subject shall not have already participated in this trial.
6. Subject specimens shall not have <10% tumor cellularity measured by H&E.
7. More than 24 months shall not have transpired between biopsy harvest and studied immunotherapy treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recurrent and metastatic Head and Neck Squamous Cell Carcinoma patients who have undergone pre-anti-PD-1/PD-L1-treatment tumor biopsy or who are scheduled for tumor biopsy prior to anti-PD-1/PD-L1 treatment will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Disease Control Rate: Inter-interval | through Final Analysis cutoff date of Dec 1, 2023
  Inequality comparison of the linearly increasing Disease Control Rate of patients assigned to OncoPrism-HNSCC quarters 1, 2, 3, and 4.

SECONDARY OUTCOMES:
Disease Control Rate: Inter-interval 2 | through Final Analysis cutoff date of Dec 1, 2023
  Inequality comparison of the Disease Control Rate of patients assigned to OncoPrism-HNSCC intervals 1 and 2 versus 3 and 4.
Sensitivity: OncoPrism-HNSCC vs PD-L1 IHC | through Final Analysis cutoff date of Dec 1, 2023
  Non-inferior comparison of the sensitivity of OncoPrism-HNSCC, using a binary threshold between intervals 2 and 3, versus PD-L1 IHC, using a binary threshold at CPS of 20.

CONTACTS AND LOCATIONS:
Locations (1):
- Curebase, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided